CLINICAL TRIAL: NCT01222390
Title: The Contour Profile® Tissue Expander in Immediate Breast Reconstruction: A Three-Dimensional Look Into Shape and Volume Changes
Brief Title: Tissue Expander Breast Reconstruction Study on Breast Volume and Shape Change
Acronym: CPX3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Principal Investigator, John Kim, Associate Professor Division of Plastic and Reconstructive Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G10-0056
Record Dates: First submitted 2010-10-13; First posted 2010-10-18 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Contour Irregularity of Reconstructed Breast
Keywords: Breast Cancer Reconstruction; Tissue Expander; 3-D Camera; Breast Reconstruction; Crescentric; Expander Profile; Fill-Volume; Lower Pole; Upper Pole; Acellular Dermis; 3-D Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contour Profile Tissue Exander (Experimental): Patients undergoing breast reconstruction using a Contour Profile Tissue Expander (CPX3).
  Interventions: Device: Contour Profile Tissue Expander

INTERVENTIONS:
Device: Contour Profile Tissue Expander — The Contour Profile Tissue Expander is a tissue expander with a greater height to width ratio than traditional tissue expanders. This increased ratio allows for greater lower pole expansion, thus creating a more natural looking, ptotic breast. Additionally, the suture tabs on the back of the expander hold the expander in place and prevent malposition and displacement.
  Other Names: CPX3

SUMMARY:
The purpose of this study is to explore the volume change and location of volume change in reconstructed breasts using the Contour Profile® tissue expander. Our purpose is also to investigate the safety of using CPX3® in tissue-expander breast reconstruction via a comparison between the complication rates that result from this study and the complication rates with the use of other tissue expander types, as reported in the literature. We also hope to demonstrate the use of 3-D imaging technology as an objective measure of upper and lower breast volume change and location of this volume change in the reconstructed breast. Finally, we intend to provide reconstructive surgeons with a scientific study that quantifies the patient satisfaction with aesthetic results of CPX3 in tissue expander-implant breast reconstruction. We hypothesize that the CPX3 tissue expander will provide more lower pole volume expansion when compared to lower pole volume expansion from round, standard tissue expanders as reported in the literature. Additionally, we hypothesize that CPX3, in combination with human acellular dermis, is less prone to complications than standard tissue expanders (again, as reported in the literature).

DETAILED DESCRIPTION:
Tissue expansion is an accepted and widely used method for breast reconstruction. A drawback in using standard tissue expanders is unwanted fullness at the upper pole and insufficient expansion at the lower pole of the breast. Round expanders can result in poor ptosis (sagging) because of unwanted upper pole fullness and are not without risk for complications[1, 2]. Anatomically-shaped expanders also have shortcomings and complications such as malposition[3-7]. A tissue expander designed to counteract upper pole fullness is necessary to achieve a more natural appearing ptotic breast with a well-defined inframammary fold (IMF)[8]. The inframammary fold is the crease below the breast where the breast meets the chest wall. Mentor's Contour Profile® (CPX3) tissue expander provides a design with a greater height to width ratio for greater lower pole expansion. It also has suture tabs on the back of the expander to hold the expander in place and prevent malposition. Another recent advancement in tissue expander breast reconstruction is the use of cadaveric-derived human acellular dermis for rapid intraoperative expansion and early projection[9-14].

The crescent-shaped expander has been studied by John YS Kim, MD in a retrospective review of 40 consecutive patients who underwent acellular dermis assisted breast reconstruction. He found the crescentric tissue expansion with acellular dermis is well tolerated with high patient and surgeon satisfaction likely due to selective lower pole expansion related to the crescent shape, as well as significant immediate expansion related to larger subpectoral pockets.

To date, no studies have been reported that investigate the lower pole expansion resulting from varying tissue expander dimensions with objective computer software[15, 16]. The advent of three-dimensional imaging technology to objectively measure lower pole expansion provides a quantitative means to study the advantages of using the CPX3® tissue expander. We propose a study that will show whether or not the CPX3® tissue expander's unique design can have an ultimate effect on the shape and location of volume change on the postoperative breast. Three-dimensional cameras also provide an advantage for assessing patients undergoing bilateral mastectomy and reconstruction who desire a reconstructive outcome that will bear some resemblance to their current breasts [15].

The 3-D imaging calculation evaluates the following parameters: absolute volume, absolute volume change, location of expansion, base width, breast projection and contour symmetry. Older methods of volume assessment would assume that the base of the breast is a flat plane. The Vectra system takes into account the curvature of the chest wall, which results in a more accurate breast volume measurement. With 3-D imaging there is no exposure to radiation[16]. Another advantage to 3-D imaging is the option to view the subject's image at any angle, 360 degrees[17]. Our study would show the postoperative results of using the CPX3® tissue expander with an objective analysis of the degree of lower-pole expansion.

This will be a prospective study. Fifteen patients will be enrolled and will receive a Contour profile tissue expander (CPX3) during their reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo unilateral or bilateral mastectomies for treatment of breast cancer with immediate tissue expander reconstruction

Exclusion Criteria:

* Patients who have had previous immediate non-expander based breast reconstruction
* Patients who have had delayed secondary flap surgery (replacing expander with autogenous tissue)
* Patients who have pacemakers and/or defibrillators which are not compatible with CPX3

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John YS Kim, MD, MA, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Hirsch EM, Seth AK, Dumanian GA, Kim JYS, Mustoe TA, Galiano RD, Fine NA. Outcomes of tissue expander/implant breast reconstruction in the setting of prereconstruction radiation. Plast Reconstr Surg. 2012 Feb;129(2):354-361. doi: 10.1097/PRS.0b013e31823ae8b1. PMID 22286418
- [Result] Mioton LM, Smetona JT, Hanwright PJ, Seth AK, Wang E, Bilimoria KY, Gaido J, Fine NA, Kim JY. Comparing thirty-day outcomes in prosthetic and autologous breast reconstruction: a multivariate analysis of 13,082 patients? J Plast Reconstr Aesthet Surg. 2013 Jul;66(7):917-25. doi: 10.1016/j.bjps.2013.03.009. Epub 2013 Apr 4. PMID 23562485
- [Result] Nahabedian MY, Galdino G. Symmetrical breast reconstruction: is there a role for three-dimensional digital photography? Plast Reconstr Surg. 2003 Nov;112(6):1582-90. doi: 10.1097/01.PRS.0000085818.54980.C4. PMID 14578788

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contour Profile Tissue Exander
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Contour Profile Tissue Exander
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14.2440)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Breast Projection
Description: The primary outcome of interest for this study was the change in breast projection from the time of maximum tissue expander fill volume, to 3 months after the tissue expander/implant exchange surgery. Upon final fill of the tissue expander, the breast has a certain projection. Once the fully expanded tissue expander is exchanged for the permanent implant, the patients' breast projection changes gradually over time. The change in breast projection is measured in percent change of projection from baseline (the time of the final, maximum expander fill) to 3 months after the tissue expander/implant exchange surgery (at which time a change in projection has occurred).
Time Frame: 1.5 years
Measure: Mean (Standard Deviation); unit: percentage loss of projection
Units Other Than Participants: breasts
Arm/Group | Contour Profile Tissue Exander
Number analyzed (Participants) | 12
Number analyzed (breasts) | 14
percentage loss of projection | 19.8205 (13.9231)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through 1 year post-operatively. This means 1 year after the tissue expander/implant exchange surgery.
Arm/Group | Contour Profile Tissue Exander
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contour Profile Tissue Exander (N=12)
Delayed wound healing of breast (Reproductive system and breast disorders) | 1 (1) — Patient had slight delayed wound healing of her right breast. This was debrided and then closed in layers with 3-0 Vicryl and 3-0 Prolene. Sterile dressings were applied. The patient tolerated the procedure well.

LIMITATIONS AND CAVEATS:
The number of subjects studied is small; projection measurements may have been subject to human error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No